# DEPARTMENT OF PSYCHIATRY

Department of Psychiatry Warneford Hospital, Warneford Lane Headington, Oxford Oxfordshire OX3 7JX



#### **Principal Investigator:**

Professor Catherine Harmer [DPhil supervisor] catherine.harmer@psych.ox.ac.uk

### **Primary Researcher:**

Andreea Raslescu [DPhil candidate] andreea.raslescu@psych.ox.ac.uk

# **PARTICIPANT CONSENT FORM**

CUREC Approval Reference: R74013/RE006

# Combined Antidepressant and Behavioural Intervention (CABIN) study

Purpose of Study: to investigate the effects of a combined antidepressant (citalopram) and behavioural activation intervention on the processing of emotional information

| | | Please initial each<br>box |
|---|---|---|
| 1 | I confirm that I have read and understand the information sheet version $\underline{2.0}$ dated $\underline{31}$ March $\underline{2022}$ for the above study. I have had the opportunity to consider the information carefully, ask questions and have had these questions answered satisfactorily. | |
| 2 | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, and without any adverse consequences or academic penalty. | |
| 3 | I have been advised about the potential risks associated with taking part in this research and have taken these into consideration before consenting to participate. | |
| 4 | I have been advised as to what I need to do for this research (especially with regard to citalopram intake) and I agree to follow the instructions given to me. | |
| 5 | To the best of my knowledge, I do not meet any of the exclusion criteria outlined in the information sheet for this research. If this changes at a later date during study participation, I agree to notify the researchers immediately. | |
| 6 | I understand that data collected during the study may be looked at by designated individuals from the University of Oxford. I give permission for these individuals to access my data. | |
| 7 | I understand who will have access to personal data (including special category data) provided, how the data will be stored and what will happen to the data at the end of the project. | |
| 8 | I agree for data collected in this study to be shared with other researchers, including those working outside of the UK and the EU, to be used in other research studies. I understand that any data shared will be anonymised so that I cannot be identified. | |

| 9 | rare circumstances in whi | ch it is judged that mysel | ictly confidential except in the<br>If or someone else is at risk of<br>ssary to an emergency would be |
|---|---|---|---|
| | communicated). | se only information nece | ssary to an emergency would be |
| 9 | I understand how this res | search will be written up and published. | |
| 10 | • | d that this project has been reviewed by, and received ethics clearance University of Oxford Central University Research Ethics Committee. | |
| 11 | I understand how to raise | e a concern or make a complaint. | |
| 12 | I agree to take part in the study. | | |
| Optional: | nal: I wish to receive a summary of results at the end of this study. | | |
| | | dd / mm / yyyy | |
| Name of Participant | | Date | Signature |
| | | dd / mm / yyyy | |
| Name of p | person taking consent | Date | Signature |